CLINICAL TRIAL: NCT01528982
Title: Susceptibility to Pathological Gambling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB12-1237
Record Dates: First submitted 2011-08-30; First posted 2012-02-08 (Estimated); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Pathological Gambling
MeSH Terms: conditions — Gambling | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Psychoeducation
- Mindfulness (Active Comparator): Mindfulness activity and psychoeducation
  Interventions: Behavioral: Mindfulness
- Cognition (Active Comparator): Cognitive training and psychoeducation
  Interventions: Behavioral: Cognition

INTERVENTIONS:
Behavioral: Mindfulness — Subjects receive mindfulness training
  Other Names: Training
  Arms: Mindfulness
Behavioral: Cognition — Subject receive cognitive training
  Other Names: Training
  Arms: Cognition

SUMMARY:
The goal of this study is to assess the risk factors for the development of pathological gambling.

DETAILED DESCRIPTION:
This study will track up to 600 young adults (ages 18 to 29) for a two-year period, collecting variables such as gambling behavior, drug and alcohol use, psychiatry and medical history, family history, impulsivity, quality of life, self-esteem, and cognition. For some individuals who meet criteria as being impulsive, they will be randomized to receive an intervention to help reduce their impulsivity.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the procedures and provide written consent
* Gambled at least 5 times in the past year
* Between the ages of 18 and 29 at intake

Exclusion Criteria:

* Inability to understand the procedures and provide written consent

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 588 (Actual)
Dates: Start 2008-11; Primary Completion 2024-06 (Actual); Study Completion 2024-06 (Actual)

PRIMARY OUTCOMES:
Structured Clinical Interview for Pathological Gambling (SCI-PG) | Up to 3 years
  The SCI-PG is a validated and reliable scale assessing the presence of DSM-IV criteria for pathological gambling. The number of criteria met for PG is added for a total score and those meeting 5 or more criteria have DSM-IV pathological gambling.
  Subjects are expected to be followed for the duration of the 3 year study.
  Diagnostic criteria for pathological gambling every 3 months for the length of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, JD, MD, MPH, Principal Investigator — University of Chicago, Department of Psychiatry
Locations (1):
- University of Chicago, Chicago, Illinois, United States